CLINICAL TRIAL: NCT04456647
Title: Parenteral Nutrition Therapy in Patients With Incurable Cancer - A Retrospective Analysis of Current Practice
Brief Title: Parenteral Nutrition Therapy in Patients With Incurable Cancer
Acronym: PATNIC
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset i Vestfold HF (Other); Sykehuset Telemark (Other Government); Haukeland University Hospital (Other); University of Bergen (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/1500
Record Dates: First submitted 2020-06-08; First posted 2020-07-02 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Neoplasms; Terminal Illness
Keywords: Parenteral nutrition; Medical Records; Palliative Care; Disease Progression
MeSH Terms: conditions — Neoplasms; Hyperphagia; Disease Progression | interventions — Parenteral Nutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parenteral nutrition
  Interventions: Other: Parenteral nutrition

INTERVENTIONS:
Other: Parenteral nutrition — Parenteral nutrition treatment in palliative care

SUMMARY:
Parenteral nutrition (PN) treatment in patients with incurable cancer is understudied and the level of evidence for clinical meaningful effects is weak. Guidelines give few specific recommendations regarding which patients with incurable cancer that should be offered PN treatment. According to the Norwegian prescription database, the use of parenteral nutrition has more than doubled in the period 2004-2015. These numbers do not separate between diagnoses and medical conditions, so the current use of medical nutrition in cancer patients in Norway is not known. The decision to initiate parenteral nutrition is taken at hospitals, whereupon the patient returns home to their respective municipalities and receives follow-up by the home care service. There are often uncertainties about the duration of treatment, as patients' clinical condition can change rapidly. One major challenge health care professionals face is to decide when to end medical nutrition therapy. Patients and relatives may experience fear that discontinuation of medical nutrition accelerates death, while health care professionals often experience that nutrition in many cases does not help and inflicts negatively on patients' condition. This makes communication concerning end of nutritional treatment between health care professionals at several health care levels, patients and their relatives challenging.

There is a need for a stronger evidence base considering the effect of medical nutrition in patients with incurable cancer. To be able to study the effect of PN treatment, more studies on clinical practice of PN treatment to patients with incurable cancer is needed. Aspects like indication for use, dosage and duration of PN treatment is poorly described in the available literature. Thus, the aim of this study is to describe indications for use of PN, duration of treatment, reasons for discontinuation, method of administration, possible benefits and complications as well as survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient with incurable cancer
* Use of parental nutrition in palliative setting

Exclusion Criteria:

* Still alive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective medical record review includes adult patients with incurable cancer who received parenteral nutrition treatment in palliative care in the time period, January 2011 to December 2017. Only patients who were deceased at point of data abstraction are included.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Received dose of parenteral nutrition | From start of parenteral nutrition treatment to termination of parenteral nutrition, up to 3 years
  Dose is measured in kcal/kg/day
Duration of treatment | From start of parenteral nutrition treatment to termination of parenteral nutrition, up to 3 years
  Duration is measured in days
Survival | From start of parenteral nutrition treatment to date of death, up to 7 years
  Survival is measured in days
Indication for use of parenteral nutrition | Baseline
  Registered indication for use of parenteral nutrition treatment

CONTACTS AND LOCATIONS:
Overall Officials: Trude Rakel Balstad, phd, Principal Investigator — Norwegian University of Science and Technology; Torstein Baade Rø, md phd, Study Director — Norwegian University of Science and Technology, IKOM; Arne Solberg, md phd, Study Director — Cancer Clinic, St. Olavs hospital, Trondheim University hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Sykehuset Telemark, Skien
  - St Olavs Hospital, Trondheim
  - Sykehuset i Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: No